CLINICAL TRIAL: NCT01237964
Title: Phase 2 Of Injectable Collagenase (Xiaflex) For Burns' Associated Contracture
Brief Title: Injectable Collagenase For Burns' Associated Contracture
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Joseph Haik, MD, Director of burn's unit, Plastic Surgery Department, Sheba Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-10-7631-JH-CTIL
Record Dates: First submitted 2010-11-03; First posted 2010-11-10 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: Burn's Associated Contracture
MeSH Terms: interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xiaflex ( Collagenase use) (Experimental): all 10 patients will be selected from out burn's clinic pool and will be injected using collagenase
  Interventions: Drug: Xiaflex (FDA approved collagenase)

INTERVENTIONS:
Drug: Xiaflex (FDA approved collagenase) — 0.58mg of collagenase will be diluted in saline and injected in 3 points surrounding the limiting contracture
  Other Names: Xiaflex( Collagenase Clostridium Histolytiucm); https://www.xiaflex.com/

SUMMARY:
A pilot experiment to test the efficiency of the enzyme Collagenase in treating contractures which result's from burn's healing process.

So far, treatment of choice in patients with burn's created movement limiting contractures, concentrated around supportive care. Patients were referred to surgical intervention only if necessary. Treatment by injecting an external enzyme is avant-garde and hasn't been done under such conditions.

This study might introduce a new kind of treatment, which can be done in ambulatory environment .This type of treatment might significantly improve patients' function and quality of life, with no need for a surgical intervention.

DETAILED DESCRIPTION:
Scientific Background:

Contracture is defined as a scar tissue that replaces the original tissue and leads to shortening and tightening of the muscle results in a range of motion limitation and deformity. Contracture creation is common in burn's healing process. The process itself involves fibrosis of the effected area including intrusion towards the deep layers of the skin, and can be described as ineffective healing process. In many cases these scars have major functional and cosmetic implications that challenges the plastic surgery departments around the world.

Creation of bands, webs and contractures close to a joint area can cause a significant movement limitation and shortens the range of motion. Until recently, failure of treatment with bandaging, splints and physiotherapy activity usually led to surgical intervention involving many kinds of techniques ranging from simple incisions, Z-Plasties to skin grafts, and flaps. All these methods were meant to release the contracture itself and restore the functional capability.

A recent study showed that it's possible to use the collagenase enzyme in releasing dupuytren's contracture by a simple injection, a procedure that can be preformed under ambulatory conditions. This kind of contracture causes a fixed flexion of the fingers towards the palm of the hand. The study was a double blinded, placebo controlled study and involved 308 patients, all suffered from contracture with at least 20 degrees range of movement limitation. In the end, it was proved beyond any doubt that collagenase is effective in releasing and restoring range of motion of dupuytren's contracture. These positive results might indicate the possibility of using collagenase in other kinds of contractures.

In this study the investigators intend to perform a preliminary test of the effectiveness of collagenase in treating contracture that developed due to the burn's healing process. As comparison parameters the investigators will compare the range of motion before and after treatment and subjective feeling of pain (again, before and after treatment) according to VAS scale of pain. Also the investigators will try to monitor any kind of side effects that might appear.

In the clinical aspect, this study might introduce the medical community with a new kind of treatment protocols and even might decrease the need for surgical intervention in these patients.

Goal:

A pilot experiment to test the efficiency of the enzyme Collagenase in treating contractures which result's from burn's healing process.

Methods:

During the study the investigators will recruit about 10 patients which suffer from a known contracture that causes movement's restriction and can be attributed to burn's healing process. These patients will have to meet the exclusion and inclusion criteria of the study.

Patients will sign an informed consent in according to the Helsinki Committee, containing the list of complications and side effects expected. Patients will go through Collagenase enzyme injections according to the protocol that was conducted in the dupuytren's study. Before performing the injections, the range of motion's limitations will be measured using goniometer and a pain scale questionnaire (VAS) will be filled by the patient. Remeasuring will be done in several time periods, after the first injection, ranging from 24 hours, a week, 14 days and 28 days.

Expected results and research significance:

So far, treatment of choice in patients with burn's created movement limiting contractures, concentrated around supportive care. Patients were referred to surgical intervention only if necessary .Treatment by injecting an external enzyme is avant-garde and hasn't been done under such conditions.

Injections attempts of various enzymes such as hyaluronidase , Collagenase and also Gelatinase are documented in the literature as therapeutic trial for Keloid and hypertrophic scars in the aesthetic aspect, were found ineffective. However, literature review found no evidence of therapeutic attempts using Collagenase in burn's healing contracture for the functional aspect. These processes are known to be fibrotic and rich with collagen deposition.

This study might introduce a new kind of treatment, which can be done in ambulatory environment .This type of treatment might significantly improve patients' function and quality of life, with no need for a surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

1. age - 18+
2. Contracture is 6 month old or more
3. Place of contracture in a flex-ext joint only (e.g knee, elbow)
4. Contracture leads to 15% decrease in joint range of movement vs anatomical range
5. Physiotherapy can no longer improve those patients condition

Exclusion Criteria:

1. Any systemic condition involving skin or soft tissue disease
2. skin disease related to elastin, collagen or keratinocytes
3. Known allergy to Clostridium Collagenase enzyme
4. Psychiatric, Prisoners, Soldiers, Pregnant women
5. Patients whom due to their home location will not be available to frequent surveillance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-04 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Increase functionality of involved joint | 24 hours after injection
  range of motion of the joint involved will be measured using Goniometer
Pain assessment | 24 hours after injection
  will be measured using VAS pain scale
Increase functionality of involved joint | 14 days after injection
  range of motion of the joint involved will be measured using Goniometer
Increase functionality of involved joint | 28 days after injection
  range of motion of the joint involved will be measured using Goniometer
Pain assessment | 14 days after injection
  will be measured using VAS pain scale
Pain assessment | 28 days after injection
  will be measured using VAS pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Hospital, Ramat Gan, Israel

REFERENCES:
- [Result] Hurst LC, Badalamente MA, Hentz VR, Hotchkiss RN, Kaplan FT, Meals RA, Smith TM, Rodzvilla J; CORD I Study Group. Injectable collagenase clostridium histolyticum for Dupuytren's contracture. N Engl J Med. 2009 Sep 3;361(10):968-79. doi: 10.1056/NEJMoa0810866. PMID 19726771
- See also: xiaflex product which will be used during the study — https://www.xiaflex.com/